CLINICAL TRIAL: NCT05299073
Title: A Randomised, Double-blind, Three-arm, Single-dose, Parallel Study to Compare the Pharmacokinetics, Pharmacodynamics, Safety, and Immunogenicity Profile of MB09 (Denosumab Biosimilar) and EU/US-sourced Xgeva® in Healthy Male Volunteers
Brief Title: A Study Comparing the Pharmacokinetic Similarity of MB09 and EU/US-Sourced Xgeva
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: mAbxience Research S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MB09-A-01-19
Record Dates: First submitted 2022-03-08; First posted 2022-03-28 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — QL1206

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MB09 (denosumab biosimilar) (Experimental): Sterile vial 120mg/1.7mL, Single dose, 35mg SC
  Interventions: Drug: MB09
- US-sourced Xgeva (Active Comparator): Sterile vial 120mg/1.7mL, Single dose, 35mg SC
  Interventions: Drug: US-sourced Xgeva
- EU-sourced Xgeva (Active Comparator): Sterile vial 120mg/1.7mL, Single dose, 35mg SC
  Interventions: Drug: EU-sourced Xgeva

INTERVENTIONS:
Drug: MB09 — Single dose of 35mg SC administered
  Other Names: denosumab biosimilar
  Arms: MB09 (denosumab biosimilar)
Drug: US-sourced Xgeva — Single dose of 35mg SC administered
  Other Names: US-licensed Xgeva
  Arms: US-sourced Xgeva
Drug: EU-sourced Xgeva — Single dose of 35mg SC administered
  Other Names: EU-licensed Xgeva
  Arms: EU-sourced Xgeva

SUMMARY:
Randomized, double blind, parallel group, single dose, 3 arm study to investigate and compare the PK, PD, safety and immunogenicity profile of MB09 with EU/US-Xgeva® in healthy male subjects.

During the course of the study, the similarity in pharmacokinetics will be assessed by sampling the levels of drug in the blood, and by comparing these levels among the different administration arms. Pharmacodynamics, safety, tolerability, and immunologic response to the administered drugs will also be evaluated throughout.

DETAILED DESCRIPTION:
The primary PK parameter endpoints are AUC0-last and Cmax for denosumab. The secondary PK endpoints will include all other PK parameters for denosumab, including AUC0-∞, Tmax, CL and t1/2.

For the primary PK Analysis, an analysis of variance (ANOVA) model with treatment and stratification factors as fixed effects will be performed on the natural log transformed values of Cmax, AUC0 last, and AUC0-∞.

Estimates of geometric mean ratios together with the corresponding 90% confidence intervals (CI) will be derived for the comparisons of the PK parameters as follows:

* MB09 versus EU-Xgeva®
* MB09 versus US-Xgeva®
* EU-Xgeva® versus US-Xgeva®

Bioequivalence will be concluded if the 90% CIs for the test to reference ratios of the geometric least square means for AUC0-last and Cmax are entirely contained within the [80%, 125%] interval.

For the PD Analysis, an analysis of covariance (ANCOVA) model with treatment and stratification factors as fixed effects and logged pre-dose sCTX concentrations fitted as a covariate will be performed on the natural log-transformed values of AUEC0 253 and AUIC0 253.

Adverse events will be coded using MedDRA Version 24. All AE data will be presented in a data listing. Treatment-emergent AEs will be summarised by treatment and overall, as well as by severity and relationship to study drug. Serious AEs and AEs leading to discontinuation of study drug will also be presented in the data listings and summarised by treatment and overall.

The incidence of ADA to denosumab and the neutralizing potential and titre of positive ADAs will be reported. All immunogenicity data will be presented in the data listings.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a male of any race, between 28 and 55 years of age, inclusive, at screening.
2. The subject has a BMI between 18.5 and 29.9 kg/m2, inclusive, (total body weight between 60 and 95 kg, inclusive) at screening and check-in.
3. The subject is considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results (congenital nonhaemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is acceptable), vital sign measurements (systolic BP ≥90 mm Hg and ≤140 mm Hg, diastolic BP ≥50 mm Hg and ≤90 mm Hg), 12 lead ECG results, and physical examination findings at screening and check in.
4. The subject must use an adequate method of contraception (eg, condom) or be willing to practice sexual abstinence during the study starting from the day of dosing and for 140 days after dosing. The subject must agree to not donating sperm during the study and for at least 140 days after dosing. Participating subject's female partner of childbearing potential should use an additional form of contraception such as an intra uterine device, barrier method with spermicide, oral contraceptive, injectable progesterone, or sub-dermal implant starting from the male partner's day of dosing until at least 140 days after dosing. The female partner of the participating subject should be familiar with the use of the respective contraceptive methods. Intra-uterine devices and hormonal methods for contraception should be used for at least 1 menstruation cycle prior to the administration of study drug.
5. The subject must be able to comprehend and willing to sign an ICF and to abide by the study restrictions. Subjects must have signed an ICF before any study-related procedure or evaluation is performed.

Exclusion Criteria:

1. The subject has had previous exposure to denosumab.
2. The subject has a significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator.
3. The subject has a history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator.
4. The subject has any current or recent history of infections, including localised infections (within 2 months prior to screening for any serious infection that requires hospitalisation or IV anti-infective or within 14 days prior to screening for any active infection which requires oral treatment).
5. The subject has a dental or jaw disease requiring oral surgery or dental surgery within 6 months prior to study product administration or plans to have dental surgery within 6 months after dosing.
6. The subject has a history of osteomyelitis or osteonecrosis of the jaw requiring suturing within 30 days before dosing, or within 30 days after the last study visit.
7. The subject has a medically significant dental disease or dental neglect, with signs and/or symptoms of local or systemic infection that would likely require a dental procedure during the course of the study. Standard dentistry treatments (eg, dental filling or prophylaxis/cleaning) are allowed.
8. The subject has clinically relevant history of alcoholism, addiction or drug/chemical abuse prior to check in, and/or positive urinary test for alcohol or drugs of abuse at screening or check in.
9. The subject has positive hepatitis panel (HBV and HCV) or positive HIV test. Subjects whose results are compatible with prior immunisation and not infection may be included at the discretion of the investigator.
10. The subject has participated in a clinical study involving administration of an investigational drug (new chemical entity), with dosing in the past 90 days prior to Day 1, or within 5 half-lives of the investigational drug used in the study, whichever is longer.
11. The subject has used or intends to use slow-release medications/products considered to still be active within 30 days prior to check in, unless deemed acceptable by the investigator.
12. The subject has used or intends to use any nonprescription medications/products (except paracetamol [up to 2 g/day] and ibuprofen [800 mg/day]), including vitamins, minerals, supplements (eg, Biotin), and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to check in, unless deemed acceptable by the investigator. Vitamin C, vitamin D, and calcium in daily recommended doses (≤1000 mg elemental calcium and 1000 IU vitamin D based on screening levels of vitamin D) are allowed.
13. The subject has received the COVID-19 vaccine within 14 days before Day 1 or plans to receive a COVID-19 vaccine within 12 weeks after study drug dosing or has positive test for COVID 19 during screening or presence of COVID 19 symptoms within 4 weeks prior to Day -1.
14. The subject has received a live or attenuated vaccine within 3 months prior to screening or has the intention to receive a vaccine during the study. The subject intends to travel to a region where a vaccination will be required due to endemic disease during the study.
15. The subject has used tobacco- or nicotine-containing products within 1 year prior to check-in or anytime during the study, or has a positive cotinine test upon screening or check-in.
16. The subject has donated blood within 60 days prior to dosing, plasma from 14 days prior to screening, or platelets from 42 days prior to dosing.
17. The subject has poor peripheral venous access.
18. Subjects who, in the opinion of the investigator, should not participate in this study.

Ages: 28 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male subjects may be enrolled
Enrollment: 257 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-18 (Actual); Study Completion 2023-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monika Tomaszewska-Kiecana, MD, Principal Investigator — Biokinetica S.A.
Locations (1):
- Biokinetica - Early Phase Institute, Józefów, Poland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MB09 (Denosumab Biosimilar): Sterile vial 120mg/1.7mL, Single dose, 35mg SC
  MB09 (denosumab biosimilar): Single dose of 35mg SC administered
Period: Overall Study
Arm/Group | MB09 (Denosumab Biosimilar) | US-sourced Xgeva | EU-sourced Xgeva
Started | 85 | 86 | 86
Completed | 85 | 84 | 85
Not Completed | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: In the EU-sourced Xgeva arm, 1 (1.2%) subject withdrew before receiving the study treatment. In the US-sourced Xgeva arm, 1 (1.2%) subject was discontinued from the study due to an AE of temperature increased, before receiving the study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | MB09 (Denosumab Biosimilar) | US-sourced Xgeva | EU-sourced Xgeva | Total
Number analyzed (Participants) | 85 | 85 | 85 | 255
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 85 | 85 | 85 | 255
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (6.93) | 38.8 (6.59) | 39.4 (7.15) | 39.5 (6.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 85 | 85 | 85 | 255
Race/Ethnicity, Customized [Number; unit: participants]
  Race & Ethnicity : White | 85 | 85 | 85 | 255
  Race & Ethnicity : Not Hispanic or Latino | 85 | 85 | 85 | 255
Region of Enrollment [Count of Participants; unit: Participants]
  Poland | 85 | 85 | 85 | 255
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.13 (2.441) | 25.76 (2.344) | 26.05 (2.415) | 25.98 (2.396)
Weight [Mean (Standard Deviation); unit: Kg] | 83.68 (8.550) | 82.74 (8.334) | 82.48 (8.643) | 82.97 (8.492)
Height [Mean (Standard Deviation); unit: cm] | 179.07 (6.098) | 179.20 (6.662) | 177.72 (5.857) | 178.66 (6.227)

OUTCOME MEASURES:

1. Primary Outcome: AUC0-last
Description: Area under the plasma concentration versus time curve from time zero to the last quantifiable concentration
Time Frame: Day 1 to Day 253
Population: Pharmacokinetic population includes subjects who received the study treatment, who did not have major protocol deviations, and had sufficient data to calculate primary PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | MB09 (Denosumab Biosimilar) | US-sourced Xgeva | EU-sourced Xgeva
Number analyzed (Participants) | 85 | 85 | 85
day*ng/mL | 146000 (26.8) | 134000 (27.4) | 138000 (24.1)

2. Primary Outcome: Cmax
Description: Maximum observed plasma concentration
Time Frame: Day 1 to Day 253
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MB09 (Denosumab Biosimilar) | US-sourced Xgeva | EU-sourced Xgeva
Number analyzed (Participants) | 85 | 85 | 85
ng/mL | 3240 (22.0) | 3100 (27.0) | 3090 (25.4)

3. Secondary Outcome: AUC0-∞
Description: Area under the plasma concentration versus time curve from time zero extrapolated to infinity
Time Frame: Day 1 to Day 253
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | MB09 (Denosumab Biosimilar) | US-sourced Xgeva | EU-sourced Xgeva
Number analyzed (Participants) | 85 | 85 | 85
day*ng/mL | 147000 (26.9) | 136000 (27.4) | 139000 (24.3)

4. Secondary Outcome: Tmax
Description: Time to reach Cmax
Time Frame: Day 1 to Day 253
Population: as for outcome 1
Measure: Median (Full Range); unit: day
Arm/Group | MB09 (Denosumab Biosimilar) | US-sourced Xgeva | EU-sourced Xgeva
Number analyzed (Participants) | 85 | 85 | 85
day | 10.00 [1.95 to 43.04] | 9.95 [3.02 to 27.99] | 9.99 [2.97 to 28.02]

5. Secondary Outcome: CL
Description: Clearance
Time Frame: Day 1 to Day 253
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | MB09 (Denosumab Biosimilar) | US-sourced Xgeva | EU-sourced Xgeva
Number analyzed (Participants) | 85 | 85 | 85
L/day | 0.238 (26.9) | 0.258 (27.4) | 0.251 (24.3)

6. Secondary Outcome: t1/2
Description: Terminal half-life
Time Frame: Day 1 to Day 253
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | MB09 (Denosumab Biosimilar) | US-sourced Xgeva | EU-sourced Xgeva
Number analyzed (Participants) | 85 | 85 | 85
days | 12.5 (38.6) | 12.1 (37.2) | 12.4 (37.6)

7. Secondary Outcome: Pharmacodynamics (sCTX) AUEC0-253
Description: Observed concentration of serum C-terminal telopeptide of Type 1 collagen (sCTX) parameter will be calculated as PD endpoint. AUC0-253: area under the plasma concentration versus time curve from time 0 to day 253
Time Frame: Day 1 to Day 253
Population: Absolute sCTX concentrations below the limit of quantification were taken as ½ lower limit of quantification (LLOQ) for parameter estimation (LLOQ: 70.0 pg/mL).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | MB09 (Denosumab Biosimilar) | US-sourced Xgeva | EU-sourced Xgeva
Number analyzed (Participants) | 85 | 85 | 85
day*ng/mL | 30000 (57.2) | 31800 (61.5) | 33400 (45.8)

8. Secondary Outcome: Incidence of Treatment Emergent Adverse Events (TEAEs)
Description: A treatment-emergent adverse event is defined as any event not present before exposure to study drug or any event already present that worsens in intensity or frequency after exposure.
Time Frame: Day 1 to Day 253
Population: At each level of subject summarization, a subject is counted once for the most related event. Percentages are based on the number of subjects in the Safety Population within each treatment and overall.
Measure: Count of Participants; unit: Participants
Arm/Group | MB09 (Denosumab Biosimilar) | US-sourced Xgeva | EU-sourced Xgeva
Number analyzed (Participants) | 85 | 85 | 85
Participants
  Any TEAE | 18 | 17 | 28
  Any Grade 1 TEAE | 4 | 3 | 5
  Any Grade 2 TEAE | 10 | 11 | 14
  Any Grade 3 or higher TEAE | 9 | 4 | 13
  Any serious TEAE | 2 | 0 | 0

9. Secondary Outcome: Incidence of Anti-denosumab Antibodies (ADA)
Description: The incidence of ADA to denosumab and the neutralizing potential and titre of positive ADA.
  The immunogenicity endpoint included denosumab anti-drug antibodies (ADA).
Time Frame: Day 1 to Day 253
Population: Treatment-induced ADA positive (TIADA): includes subjects with only post-treatment positive ADA results.
  Overall: includes all subjects with any TIADA positive result at any time. Percentages are based on TIADA positive subjects in the Safety population within each treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MB09 (Denosumab Biosimilar) | US-sourced Xgeva | EU-sourced Xgeva
Number analyzed (Participants) | 84 | 84 | 84
Participants
  overall negative ADA | 83 | 83 | 82
  overall positive ADA | 1 | 1 | 2

10. Secondary Outcome: Incidence of Neutralizing Antibodies (NAb)
Description: The incidence the neutralizing potential and titre of positive ADA.
Time Frame: Day 1 to Day 253
Measure: Count of Participants; unit: Participants
Arm/Group | MB09 (Denosumab Biosimilar) | US-sourced Xgeva | EU-sourced Xgeva
Number analyzed (Participants) | 85 | 85 | 85
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events and SAEs were assessed for 36 weeks (during the duration of the study) and followed until they were resolved, stable, or judged by the investigator to be not clinically significant.
Arm/Group | MB09 (Denosumab Biosimilar) | US-sourced Xgeva | EU-sourced Xgeva
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/85 | 0/85
Serious Adverse Events (participants affected / at risk) | 2/85 | 0/85 | 0/85
Other Adverse Events (participants affected / at risk) | 18/85 | 17/85 | 28/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MB09 (Denosumab Biosimilar) (N=85) | US-sourced Xgeva (N=85) | EU-sourced Xgeva (N=85)
Serious Adverse Event (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — Grade 3 SAE of osteoma
Serious Adverse Event (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Grade 3 SAE of Depression
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MB09 (Denosumab Biosimilar) (N=85) | US-sourced Xgeva (N=85) | EU-sourced Xgeva (N=85)
TEAE (Investigations) | 7 (10) | 3 (3) | 12 (16)
TEAE (Infections and infestations) | 6 (6) | 6 (9) | 6 (6)
TEAE (Nervous system disorders) | 3 (4) | 2 (2) | 3 (3)
TEAE (Injury, poisoning and procedural complications) | 1 (2) | 2 (2) | 3 (3)
TEAE (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (5)
TEAE (Gastrointestinal disorders) | 1 (1) | 1 (3) | 0 (0)
TEAE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
TEAE (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1)
TEAE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
TEAE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
TEAE (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
TEAE (General disorders) | 0 (0) | 0 (0) | 1 (1)
TEAE (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
TEAE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
TEAE (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Treatment-Related TEAE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Treatment-Related TEAE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Treatment-Related TEAE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT05299073/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-04): https://cdn.clinicaltrials.gov/large-docs/73/NCT05299073/SAP_001.pdf